CLINICAL TRIAL: NCT00421902
Title: Acupuncture Treatment for Hot Flashes in Men With Prostate Cancer, A Phase I/II Study
Brief Title: Acupuncture Treatment for Hot Flashes Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Presbyterian Brooklyn Methodist Hospital (Other)
Responsible Party: Principal Investigator, Hani Ashamalla, MD, Chairman of Radiation Oncology Department, New York Presbyterian Brooklyn Methodist Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYM # 325
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Prostate Cancer
Keywords: Hot flashes, prostate cancer, acupuncture
MeSH Terms: conditions — Prostatic Neoplasms; Hot Flashes | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Acupuncture to pevent hot flushes

ARMS (1):
- Acupuncture (Experimental): Acupuncture of the patients
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Patients will be have acupuncture (with electro stimulation)

SUMMARY:
Patients with prostate cancer who are / were treated with hormonal treatment and developed hot flashes as a side effect are offered Acupuncture as an investigational intervention. The treatment is performed twice a week for four weeks, then once a week for the following six weeks

DETAILED DESCRIPTION:
Patients with prostate cancer who are / were treated with hormonal treatment and developed hot flashes as a side effect are offered Acupuncture as an investigational intervention. The treatment is performed twice a week for four weeks, then once a week for the following six weeks. Acupuncture was done according to specific guidelines and mapping.

ELIGIBILITY:
Inclusion Criteria:

* Treatment for prostate cancer using hormonal ablation therapy
* Average of three or more hot flashes a day
* Performance Status (Karnofsky ≥ 60)
* Patients must be ≥ 18 years of age
* No other clinically significant disease
* Signed study-specific consent form prior to study entry

Exclusion Criteria:

* Initiation of a new chemotherapy regimen, immunotherapy; or initiation/ cessation of hormonal therapy during the study or for 3 weeks before the start of the study
* Pharmacological treatment of hot flashes or use of selective serotonin reuptake inhibitors (unless the dose and patients' condition have been stable for 4 weeks)
* Skin infections
* Patients who had acupuncture treatment in the 6 weeks prior to entering the study, or acupuncture given specifically for the treatment of hot flashes in the previous 6 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Relief from the hot flashes as determined by the hot flashes scoring system. | 6 months
  A Questionnaire was given to the patients to determine the relief of hot flashes

CONTACTS AND LOCATIONS:
Overall Officials: Hani Ashamalla, MD, FCCP, Principal Investigator — NY Methodist Hospital
Locations (1):
- NYP- Brooklyn Methodist Hospital, Brooklyn, New York, United States

REFERENCES:
- [Derived] Ashamalla H, Jiang ML, Guirguis A, Peluso F, Ashamalla M. Acupuncture for the alleviation of hot flashes in men treated with androgen ablation therapy. Int J Radiat Oncol Biol Phys. 2011 Apr 1;79(5):1358-63. doi: 10.1016/j.ijrobp.2010.01.025. Epub 2010 Jun 3. PMID 20605360